CLINICAL TRIAL: NCT05622201
Title: A Randomized Controlled Trial With Rituximab for Psychotic Disorder in Adults
Acronym: RCT-RITS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 278825
Record Dates: First submitted 2022-11-14; First posted 2022-11-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: RCT; immunomodulatory treatment; psychosis; rituximab; CD20 antibodies
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Psychotic Disorders | interventions — Rituximab; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A proof-of-concept study: a multicenter, placebo-controlled, double-blinded, add-on intervention study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rituximab (Experimental): Rituximab 1000 mg, infusion
  Interventions: Drug: Rituximab
- Placebo (Placebo Comparator): Saline infusion
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Infusion
  Other Names: Saline

SUMMARY:
Immunological factors are assumed to be determinants for some psychiatric disorders, thus anti-inflammatory drugs may be helpful. However, studies on such treatments are scarce. An inflammatory modulating drug rituximab, cluster of differentiation antigen 20 antibodies (anti-CD20 antibodies), is a standard treatment for e.g. multiple sclerosis.

The investigators aim to test rituximab in a randomised placebo-controlled double-blinded, add-on treatment trial in 120 participants (18-55 years) with schizophrenia spectrum disorder. Sampling from blood for analyses of inflammatory mediators are investigated at gene and protein levels and resting state functional magnetic resonance imaging (rsfMRI) and lumbar puncture are optional. Biomarkers will be investigated in relation to treatment response.

Family member(s) to the patient and the patient (separate) will be asked to participate in a qualitative interview by an independent researcher after 3 months.

DETAILED DESCRIPTION:
Immunological factors are assumed to be determinants for some psychiatric disorders, thus anti-inflammatory drugs may be helpful. However, studies on such treatments are scarce. Rituximab (anti-CD20 antibodies), a standard treatment for multiple sclerosis in Sweden, is an inflammatory modulating drug. In a small open pilot trial, markedly ill, treatment-resistant participants with schizophrenia spectrum disorder were treated with a single- dose rituximab (1000 mg), as add-on treatment to antipsychotics in Örebro, Sweden (2019-2022). Large improvements in all types of psychotic symptoms were evident, with long-lasting effects and few side-effects in most of the participants.

This is a proof-of-concept study based on our earlier findings. The investigators will conduct a multicenter, placebo-controlled, double-blinded, add-on intervention study for 120 participants with schizophrenia spectrum disorder (18-55 years). Sampling from blood for analyses of inflammatory mediators are investigated at gene and protein levels and rsfMRI and lumbar puncture are optional at baseline and endpoints. Biomarkers will be investigated in relation to treatment response.

Participants are assessed at five time-points; week 0, 2, 7, 12 (endpoint I) and 24 (endpoint II).

Research questions:

I Does the addition of rituximab to standard psychiatric treatment improve psychotic symptoms in SSD?

II Does overall disability improve with the addition of rituximab?

III Are clinical or biological markers related to treatment response?

IV Is rituximab safe and well tolerated by participants with SSD?

V Is rituximab effective for treatment resistant SSD?

In addition family member(s) to the patient will be asked to participate in a qualitative interview by a researcher after 3 months on changes in the patient's mood and anxiety level, general functioning, behaviours, energy level, psychotic symptoms, motivation, emotional reciprocity and insight to enable a qualitative analysis. We will also ask them about their general thoughts on the study. In addition we will interview the patient after 3 months using qualitative methods.

We also aim study changes in negative symptoms with the Motivation and pleasure- self report (MAP-SR) in addition to the Positive and Negative Syndrome Scale (PANSS) scale and Self-evaluation of Negative Symptoms (SNS). Childhood onset neuropsychiatric symptoms will be investigated retrospectively by the use of Five-to-Fifteen Brief (FTF-Brief).

ELIGIBILITY:
Inclusion Criteria:

1. ages 18 to 55 years
2. duration of illness exceeding 1 year
3. diagnosed with Schizophrenia spectrum disorder (SSD) according to The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
4. if female and with any risk for pregnancy, willing to use contraceptives or abstinence if normal and preferred lifestyle.
5. participants should be judged by the investigator to be lucid and oriented to person, place, time, and situation when giving the informed consent.
6. insufficiently recovered from previous antipsychotic treatments.
7. a minimum score of 4 (moderately ill) in Clinical global impression - severity (CGI-S) at baseline.

Exclusion Criteria:

1. pregnancy or breast-feeding
2. weight below 40 kg
3. clinically relevant ongoing infection at the discretion of the physician
4. chronic infections
5. positive test for hepatitis B, hepatitis C, HIV, or tuberculosis
6. malignancy currently or within 2 years prior to inclusion
7. current severe heart failure (NYHA grade IV) or any other severe heart disease (e.g. or history of cardiac arrhythmia or myocardial infarction)
8. any change of antipsychotic medication within the previous 4 weeks
9. unable to make an informed decision to consent to the trial
10. ongoing clozapine treatment
11. ongoing immunomodulatory treatment
12. treatments with monoclonal antibodies within 1 year before the inclusion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders to treatment, rated as much or very much improved with CGI-I | Baseline up to week 12
  Improvement according to clinical rated Clinical Global Impression-Improvement (CGI-I)

SECONDARY OUTCOMES:
Improvement in functioning | Baseline up to week 12 and 24
  Measuring overall disability with Personal and Social Performance Scale (PSP)
Change in psychotic symptoms | Baseline up to 12 weeks
  Change in scores in the measure for psychotic symptoms "the Positive and Negative Syndrome Scale (PANSS)"
Proportion of responders to treatment, rated as much or very much improved with CGI-I | Baseline up to week 24
  Improvement according to clinical rated Clinical Global Impression-Improvement (CGI-I)
Improvement since baseline | Baseline up to week 12 and 24
  Improvement according to clinical rated Clinical Global Impression-Improvement (CGI-I)
Change in severity since baseline | Baseline up to week 12 and 24
  Improvement according to clinical rated Clinical Global Impression-Severity (CGI-S)
Improvement in psychotic symptoms since baseline | Baseline up to week 24
  Change in scores in the measure for psychotic symptoms "the Positive and Negative Syndrome Scale (PANSS)".
Change in self-rated overall health | Baseline up to week 12 and 24
  Differences in patient self-rated health (VAS-health)
Patient-rated improvement | Baseline up to week 12 and 24
  Patient's Global Evaluation of improvement (PGE) corresponding to the CGI-I scores
Inflammatory markers in blood and/or cerebro spinal fluid (CSF) | Baseline up to week 12 and 24
  Baseline levels of inflammatory markers in relation to treatment response (optional)
Safety and tolerability of rituximab | Baseline up to week 12 and 24
  Open questions and a questionnaire (AAR-Revised)
fMRI | Baseline up to week 12 and 24
  Change in brain morphology and/or activity in fMRI (optional)
Patient-rated change in psychiatric symptoms | Baseline up to week 12 and 24
  Mental health symptom domains (Level 1 Cross-cutting symptom measure of global symptom severity) in relationship to response.

OTHER OUTCOMES:
Depression | Baseline up to week 12 and 24
  The depression item A6 in PANSS will be investigated separately
Negative symptoms | Baseline week 12 and week 24
  The Negative Syndrome Scale assessed by the clinician will be compared to self-rated negative symptoms measured with the Motivation and pleasure- self report (MAP-SR) in order to study how well they are correlated.
Qualitative assessment | 12-18 weeks after infusion
  An informant will be interviewed on whether they can see changes in patients and patient will be interviewed separately on symptoms after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Bejerot, MD, PhD, Principal Investigator — Region Örebro län
Locations (1):
- Örebro university hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bejerot S, Eklund D, Hesser H, Hietala MA, Kariis T, Lange N, Lebedev A, Montgomery S, Nordenskjold A, Petrovic P, Soderbergh A, Thunberg P, Wikstrom S, Humble MB; RCT-Rits study collaboration group. Study protocol for a randomized controlled trial with rituximab for psychotic disorder in adults (RCT-Rits). BMC Psychiatry. 2023 Oct 23;23(1):771. doi: 10.1186/s12888-023-05250-5. PMID 37872497

DOCUMENTS (1):
  • Informed Consent Form (2023-08-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT05622201/ICF_000.pdf